CLINICAL TRIAL: NCT02962232
Title: Evaluation the Safety and Efficacy of the Paclitaxel Releasing Peripheral Balloon Dilatation Catheter （LEGFLOW）in Treatment of Stenosis or Occlusion in Below The Knee Arteries: A Prospective, Multicenter, Randomized, Controlled Clinical Study
Brief Title: A Study of Below The Knee Arteries' Stenosis or Occlusion Treated With LEGFLOW OTW
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ZhuHai Cardionovum Medical Device Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LEGFLOW-2015-02
Record Dates: First submitted 2016-11-07; First posted 2016-11-11 (Estimated); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Peripheral Artery Disease
Keywords: drug eluting balloon; arterial vasculature below the knee
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LEGFLOW OTW group (Experimental): in the LEGFLOW OTW group the subject will be treated by the Paclitaxel Releasing Peripheral Balloon Dilatation Catheter (LEGFLOW)
  Interventions: Device: Paclitaxel Releasing Peripheral Balloon Dilatation Catheter
- AMPHIRION DEEP group (Active Comparator): in the AMPHIRION DEEP group the subject will be treated by PTA catheter (AMPHIRION DEEP)
  Interventions: Device: PTA catheter

INTERVENTIONS:
Device: Paclitaxel Releasing Peripheral Balloon Dilatation Catheter — treatment group
  Other Names: LEGFLOW OTW
  Arms: LEGFLOW OTW group
Device: PTA catheter — control group
  Other Names: AMPHIRION DEEP
  Arms: AMPHIRION DEEP group

SUMMARY:
To evaluate the safety and efficacy of the Paclitaxel Releasing Peripheral Balloon Dilatation Catheter (LEGFLOW) compared to the PTA catheter (AMPHIRION DEEP) in treatment of stenosis or occlusion in below the knee artery.

DETAILED DESCRIPTION:
To evaluate the safety and efficacy of the Paclitaxel Releasing Peripheral Balloon Dilatation Catheter (LEGFLOW) compared to the PTA catheter (AMPHIRION DEEP) in treatment of stenosis or occlusion inbelow the knee artery.

This is a prospective, multi-center, randomized, control, opening, superiority designed clinical study. Plan to enroll 172 eligible subjects in 15 centers in China, all these subjects will be randomized 1:1 to the study group (LEGFLOW OTW group, n=86) and control group (AMPHIRION DEEP group, n=86), and accept the treatment of LEGFLOW OTW and AMPHIRION DEEP respectively.

ELIGIBILITY:
Inclusion Criteria:

* age from 18 to 85 years (include 18 and 85 year);
* critical limb ischemia subjects (Rutherford classification from 3 to 6)
* expective survival more than 1 year;
* can understand the study objective, self willing enrolls and sign the informed consent, and accept scheduled followed up at the specific time.

Angiographic inclusive criteria:

* reference vessel diameter 2.0-3.5mm;
* stenosis or occlusion in arterial vasculature below the knee shall have distal outflow;
* target lesion stenosis ≥70% or occlusion, length ≤270mm;
* if subject has ipsilateral / contralateral iliac lesions, the iliac lesion shall meet all the following criteria:

  * iliac lesion or occlusion length ≤100mm and
  * shall be treated earlier than the target lesion and
  * shall be treated successfully. the successful treatment standard: 1) residual stenosis <30%; 2) without flow limiting dissection 3) without thrombosis, embolism or any other serious adverse events

Exclusion Criteria:

* subjects currently participate in other drugs or medical devices clinical study and have not reach the primary endpoint;
* childbearing aged women whose pregnancy test before intervention operation is not negative, and lactating mothers;
* subjects with renal function insufficiency (serum creatinine> 2.5mg / dL or in renal dialysis);
* subjects have known be allergy or contraindication to the contrast agent, paclitaxel, heparin, antiplatelet, anticoagulant or thrombolytic agents;
* subjects plan to a major amputation (over metatarsal level);
* stroke subjects within 3 months or stroke subjects with severe hemiplegia and aphasia associated sequelaes over 3 months before the intervention operation;
* subjects with acute myocardial infarction, thrombolytic therapy or angina within 30 days before the intervention operation;
* subjects whose target lesion limb have gangrene (the gangrene range over the metatarsophalangeal joint);
* target lesion is a stenosis or occlusion that have prior been treated by scaffold implantation, DEB, ordinary balloon catheter or bypass graft;
* lesions and /or occlusion locate or extend to popliteal artery or below ankle joint;
* subjects requiring be intervention in bilateral lower limb;
* the stenosis lesion of ipsilateral femoral artery or ipsilateral popliteal artery have a diameter stenosis ≥50% untreated before the intervention operation;
* ipsilateral femoral artery or ipsilateral popliteal artery has single or adjacent lesion length ≥15cm, or ipsilateral femoral artery or ipsilateral popliteal artery has multiple lesion and one of these multiple lesion length ≥10cm or occlusion;
* - adjacent lesion: 1) interval no more than 30 mm, 2) can be treated as a single lesion;
* - multiple lesion: 1) interval no more than 30 mm, 2) need to be treated as multiple lesion;
* the residual stenosis still ≥30%, even when the length <15cm and stenosis ≥50% single or adjacent lesion in ipsilateral femoral artery or ipsilateral popliteal artery has been treated, or when each lesion length <10cm and stenosis ≥50% multiple lesion in ipsilateral femoral artery or ipsilateral popliteal artery has been treated;
* DES and /or DEB has been used in the inflow vessel of lesions treatment;
* subject has no patency vessel below the ankle artery before the intervention operation;
* target vessel aneurysm;
* acute or subacute thrombosis in target vessel;
* angiography shows severe calcification in the target lesion (before contrast injection or digital subtraction angiography, intensive annular calcifications that make target lesion not expansion and / or a calcification within the target lesion and locate on either sides of the vessel wall whose continuous length over than 5cm);
* lesions that the guild wire cannot pass through;
* subjects need be treated by thrombus endarterectomy, percutaneous transluminal plaque circumcision or laser treatment device indicate by intraoperative angiography;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2016-11; Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Target lesion restenosis determined by CTA | 6 month post procedure
  Restenosis defined as within the ± 5mm range beyond proximal and / or distal of target lesion, the lumen loss is greater than 50% of the reference vessel lumen diameter (RVD) follow-up by CTA.
  Target lesion revascularization (TLR): clinical symptoms of peripheral arterial disease recurrence or worsening, and any target lesion re-intervention caused by diameter stenosis ≥50% (confirmed by Doppler ultrasound, DSA or CT angiography).

SECONDARY OUTCOMES:
device success rate | at 0-30 days
  device success defines as: the device successfully delivered to the target location, inflated, deflated and withdrawn from the treated balloon inflation tube.
operation success rate | at 0-30 days
  operation success defines as: the blood supply of the target lesion regained after treatment, residual stenosis less than 50% and without flow-limiting dissection (≥type D) occurred.
clinical success rate | at 0-30 days
  clinical success defines as: operation success, and without any postoperative complication before discharge (death, lesions limb amputation, target lesion thrombosis or TVR)
change of the Rutherford score | in day 0-30, 6th month, 12th month post operation
change of the life equality by EQ5D | in day 0-30, 6th month, 12th month post operation compares to baseline
target limb ulcer healing rate | in day 0-30, 6th month, 12th month post operation
  healing or not, if not: improve, no change, or progression;
target lesion revascularization rate | in day 0-30, 6th month, 12th month post operation
target limb upper amputation and lower amputation rate | in day 0-30, 6th month, 12th month post operation
major adverse event rate including all cause death, target limb upper amputation and target lesion revascularization | in day 0-30, 6th month, 12th month post operation

CONTACTS AND LOCATIONS:
Overall Officials: Chen zhong, professor, Principal Investigator — Beijing Anzhen Hospital
Locations (19):
- China (19):
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Hainan General Hospital, Haikou, Hainan
  - Hebei General Hospital, Shijiazhuang, Hebei
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Beijing Anzhen Hospital Capital Medical University, Beijing
  - Beijing Chao-Yang Hospital, Beijing
  - Beijing Frendship Hospital, Capital Medical University, Beijing
  - Beijing Hospital, Beijing
  - Beijing Shijitan Hospital, Capital Medical University, Beijing
  - Chinese PLA General Hospital, Beijing
  - Fuwai Hospital, Chinese Accadamy of Medical Sciences, Beijing
  - Renji Hospital Shanghai Jiaotong University School of Medicine, Shanghai
  - Shanghai Ninth people's Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Tianjing Medical University General Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: Undecided